CLINICAL TRIAL: NCT00513682
Title: Efficacy and Safety of Ultrase® MT20 in Improving the Coefficient of Fat Absorption (CFA%) in Children With Cystic Fibrosis (CF) and Pancreatic Insufficiency (PI)
Brief Title: Efficacy and Safety of Ultrase® MT20 in Improving the Coefficient of Fat Absorption (CFA) in Children With Cystic Fibrosis (CF) and Pancreatic Insufficiency (PI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMT20CF07-01
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Pancreatic insufficiency; Steatorrhea; Children 7 to 11 years; Pancreatic enzyme
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Steatorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrase® MT20 (Experimental)
  Interventions: Drug: Ultrase® MT20

INTERVENTIONS:
Drug: Ultrase® MT20 — Ultrase® MT20 capsules will be administered orally with each meal during Day 1 to 15 in screening phase at a dose based on investigator's discretion. During Day 12 to 15, participants will receive high-fat diet and Ultrase® MT20 dose will be adjusted depending on symptoms of steatorrhea. This will be followed by a washout phase of 6 to 7 days, in which participants will receive only high-fat diet; then stabilized dose of Ultrase® MT20 capsule (as identified during screening phase) will be administered orally for 7 to 11 days during treatment phase. The stabilized dose should not to exceed 2500 lipase units per kilogram body weight per meal (lipase units/kg/meal).

SUMMARY:
This is a Phase III, multicenter, open-label study, that will evaluate the improvement of nutrient absorption when participants will receive Ultrase® MT20. This study is sponsored by Aptalis (formerly Axcan). This study is performed in children from 7 to 11 years old.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, open-label study, which will quantify the improvement of nutrient absorption when participants are receiving Ultrase® MT20. The improvement will be demonstrated by comparing the CFA percent (%) and CNA% obtained during a washout of enzyme with the CFA% and CNA% obtained during a period of treatment with Ultrase® MT20. The study is also designed to obtain safety data in CF children suffering also from PI taking Ultrase® MT20. The total duration for the participation of children in this study will be approximately up to 38 days and will include 3 phases: screening phase, the washout phase and treatment phase.

Screening phase: this phase will last 15 days and all participants will take Ultrase® MT20 as per investigator's discretion during this period. During the last 4 days, participants will be stabilized on a high fat diet and with Ultrase® MT20. The individual 'stabilized dose' of Ultrase® MT20 capsules will be determined for each participant based on the average number of capsules of Ultrase® MT20 taken during last 4 days.

Washout phase: this phase will last 6 to 7 days. The participants will continue the high-fat diet but will refrain from taking Ultrase® MT20 or any other enzymes. A 72-hour stool collection will be performed and all food consumed by the participants will be recorded to assess the CFA% and CNA%.

Treatment phase: this phase will last 7 to 11 days. The participants will continue the high-fat diet and will take the 'stabilized dose' of Ultrase® MT20 established during screening. Another 72-hour stool collection will be performed and all food consumed by the participants will be recorded to assess the CFA% and CNA%.

ELIGIBILITY:
Inclusion Criteria:

* After a full explanation of the study, participants or their legally authorized representative must have signed the informed consent or assent form along with a parental form
* Participants must have a confirmed diagnosis of CF based on one or more clinical features consistent with the CF phenotype, and one of the following:

  * A genotype with two identifiable mutations consistent with CF
  * A sweat chloride test greater that 60 millimole per liter (mmol/L) by quantitative pilocarpine iontophoresis
* Participants must have PI as demonstrated by a fecal elastase-1 (FE-1) concentration less than 100 microgram per gram (mcg/g) of stools (ScheBo test) and requiring pancreatic enzyme supplementation
* Participants must be clinically stable according to the physician's judgment by:

  * Medical and medication history
  * Baseline physical examination including vital signs and laboratory analyses
* Participants must be 7 to 11 years of age
* Participants must have an adequate nutritional status based on body mass index (BMI) greater than or equal to fifth percentile
* Participants must be on an optimal clinical dose of pancreatic enzymes (Ultrase® MT12 , MT18 or MT20 or other pancreatic enzyme preparations) prior to entry in the study and must tolerate this medication in the opinion of the investigator
* Participants must be able to be able to swallow capsules and eat a high-fat diet calculated as 2 gram fat per kilogram (g fat/kg) of body weight per day
* Participants must be, in the opinion of the investigator, able and willing to complete the study
* Female participants should be premenarcheal. Otherwise, a female participant of childbearing potential (WOCBP) must not be pregnant and must have practiced an acceptable method of contraception for at least 1 month prior to the study entry

Exclusion Criteria:

* Participants with a known contraindication, sensitivity or hypersensitivity to Ultrase® MT20 or any porcine protein
* Participants with a known allergy to the food, drug and cosmetic (FD&C) Blue No. 2 dye indicator (stool marker)
* Participants who are not willing to stop the prohibited medications or products at study entry and throughout the study
* Participants who use narcotics chronically and bowel stimulants and/or laxatives on a regular basis
* Participants with acute pancreatitis or acute exacerbation of chronic pancreatic disease
* Participants with an acute pulmonary infection
* Participants with a history of bowel resection
* Participants suffering from any dysmotility disorders
* Participants with chronic or severe abdominal pain
* Participants receiving enteral tube feeding and not willing to stop during the course of the study
* Participants with a significant medical disease that would compromise their welfare or confound the study results
* Participants with a history of or a current diagnosis of clinically significant portal hypertension
* Participants who have a condition known to increase fecal fat loss including celiac's disease, biliary cancer, biliary stricture, cholelithiasis, Crohn's disease, ulcerative colitis, pancreas cancer, radiation enteritis, tropical sprue, Whipple's disease, lactose intolerance, pseudomembranous colitis
* Participants with a current diagnosis or a history of complete distal intestinal obstruction syndrome (DIOS) in the past 6 months; or, participants who had 2 or more episodes of DIOS in the past year
* Participants with poorly controlled diabetes according to the investigator's opinion
* Female participants who are pregnant or lactating
* Participants who received an investigational drug within 30 days prior to entry into the study

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (3):
- United States (3):
  - University of Michigan Health System Cystic Fibrosis Center, Ann Arbor, Michigan
  - Cystic Fibrosis Center Rainbow Babies and Children's HospitalDivision, Cleveland, Ohio
  - Pennsylvania State University And the Milton S. Hershey Medical Center, Hershey, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrase® MT20: Ultrase® MT20 capsules orally with each meal during Day 1 to 15 in screening phase at a dose based on investigator's discretion. During Day 12 to 15, participants received high-fat diet and Ultrase® MT20 dose was adjusted depending on symptoms of steatorrhea. This was followed by a washout phase of 6 to 7 days, in which participants received only high-fat diet. Then the treatment phase was started which consisted of a stabilized dose of Ultrase® MT20 capsule (as identified during screening phase) orally for 7 to 11 days. The stabilized dose not to exceed 2500 lipase units per kilogram body weight per meal (lipase units/kg/meal).
Period: Screening Phase
Arm/Group | Ultrase® MT20
Started | 9
Completed | 9
Not Completed | 0
Period: Washout Phase
Arm/Group | Ultrase® MT20
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 2
Period: Treatment Phase
Arm/Group | Ultrase® MT20
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all the participants who were enrolled in the study.
Arm/Group | Ultrase® MT20
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA)
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined by the stools collected during the 72-hour period in either washout phase or treatment phase. Mean percent CFA was calculated for Day 3 to Day 5 or Day 6 of the respective phase.
Time Frame: Day 3 to Day 5 or Day 6 during washout phase and treatment phase
Population: Intent-to-treat (ITT) population included all the participants who took at least 1 dose of Ultrase® MT20 and had completed at least 1 phase (washout or treatment phase) evaluating primary and secondary efficacy parameters.
Measure: Mean (Standard Deviation); unit: Percent CFA
Groups:
- Ultrase® MT20 Washout Phase: Ultrase® MT20 capsules orally with each meal during Day 1 to 15 in screening phase at a dose based on investigator's discretion. During Day 12 to 15, participants received high-fat diet and Ultrase® MT20 dose was adjusted depending on symptoms of steatorrhea. This was followed by a washout phase of 6 to 7 days, in which participants received only high-fat diet.
- Ultrase® MT20 Treatment Phase: Participants who received Ultrase® MT20 capsules orally in screening phase and underwent washout phase, received stabilized dose of Ultrase® MT20 capsule (as identified during screening phase) orally for 7 to 11 days during treatment phase. The stabilized dose not to exceed 2500 lipase units per kilogram body weight per meal (unit/kg/meal).
Arm/Group | Ultrase® MT20 Washout Phase | Ultrase® MT20 Treatment Phase
Number analyzed (Participants) | 7 | 7
Percent CFA | 34.5 (21.35) | 82.7 (13.25)
Statistical Analysis 1: Comparison: Ultrase® MT20 Washout Phase vs Ultrase® MT20 Treatment Phase; Test type: Superiority or Other; p = 0.0013, t-test, 1 sided

2. Secondary Outcome: Percent Coefficient of Nitrogen Absorption (CNA)
Description: Percent CNA was calculated as [(nitrogen intake-nitrogen excretion)/nitrogen intake]*100, determined by the stools collected during the 72- hour period in either washout phase or treatment phase. Nitrogen intake was calculated as protein intake/6.25. Nitrogen excretion was measured as total fecal nitrogen. Mean percent CNA was calculated for Day 3 to Day 5 or Day 6 of the respective phase.
Time Frame: Day 3 to Day 5 or Day 6 during washout phase and treatment phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent CNA
Arm/Group | Ultrase® MT20 Washout Phase | Ultrase® MT20 Treatment Phase
Number analyzed (Participants) | 7 | 7
Percent CNA | 33.4 (20.06) | 79.5 (10.56)
Statistical Analysis 1: Comparison: Ultrase® MT20 Washout Phase vs Ultrase® MT20 Treatment Phase; Test type: Superiority or Other; p = 0.0009, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Day 1 of screening phase up to follow up (7 to 10 days post-treatment phase)
Description: Safety population included all participants who signed the informed consent form and took at least 1 dose of the study medication, including medication dispensed for the screening phase. Number of participants evaluable for each reporting group were 9 and 7 respectively.
Groups:
- Ultrase® MT20 Screening Phase: Ultrase® MT20 capsules orally with each meal during Day 1 to 15 in screening phase at a dose based on investigator's discretion. During Day 12 to 15, participants received high-fat diet and Ultrase® MT20 dose was adjusted depending on symptoms of steatorrhea.
- Ultrase® MT20 Washout Phase: Participants who received Ultrase® MT20 capsules orally in screening phase and underwent a washout phase, of 6 to 7 days, in which participants received only high-fat diet and refrained from taking Ultrase® MT20.
Arm/Group | Ultrase® MT20 Screening Phase | Ultrase® MT20 Washout Phase | Ultrase® MT20 Treatment Phase
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 2/9 | 6/9 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrase® MT20 Screening Phase (N=9) | Ultrase® MT20 Washout Phase (N=9) | Ultrase® MT20 Treatment Phase (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions may vary in accordance with each agreement that is negotiated with individual investigators. Sponsor will allow publication after multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and defer publication for period of time to allow Sponsor to obtain patent or other intellectual property right protection.